CLINICAL TRIAL: NCT02429011
Title: Functional MRI Studies of Emotion in Depression and Rapid Antidepressant Response
Brief Title: MRI Studies of Emotion in Depression
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James Murrough, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 10-1385; 5K23MH094707 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
Keywords: depression; MRI; treatment-resistant; imaging; ketamine
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDD: patients with current MDD
- Healthy Control (HC): healthy control volunteers

SUMMARY:
The purpose of this study is to research the effects of ketamine on brain function in patients with Major Depressive Disorder (MDD). This study is an ancillary MRI neuroimaging study being conducted in patients with MDD who are enrolled in a separate clinical trial. Healthy control volunteers are also enrolled. No drug or other intervention is given as part of this protocol per se.

To study brain activity related to emotion, the study team will use a technology called functional MRI (fMRI), which is a method for evaluating the flow of blood in the brain using a powerful magnet. fMRI does not involve exposure to radiation.

Patients will be shown a sample of images on a computer screen designed to bring about an emotional reaction. The MRI machine will then take a number of pictures of your head. By computer analysis, this machine is able to create a picture of your brain's activity. There are several tasks during scanning that involve looking at various images that represent different emotions, and the study team will be monitoring brain activity during these tasks.

Patients will be scanned before and 24 hours after receiving ketamine (as part of a separate study) to analyze treatments effects. These scans are compared to depressed patients who did not receive ketamine, as well as to healthy controls.

DETAILED DESCRIPTION:
Specific Aim 1: To characterize the function of basic neural systems involved in emotion perception and regulation in TRD.

* Experiment 1.1: Neural responses to emotional faces in TRD (neutral, low and high intensity sad facial expressions).

  o Hypothesis 1.1: Patients with TRD, relative to HC participants, will evidence increased activation in the amygdala/parahippocampal gyrus to sad compared to neutral faces.
* Experiment 1.2: Neural responses during negative emotion regulation in TRD (cognitive reappraisal).

  * Hypothesis 1.2: Patients with TRD, relative to HC participants, will show enhanced activation of the amygdala during the generation of negative affect and will be impaired in their ability to recruit PFC/ACC regions during attempts to down-regulate negative affect.

Specific Aim 2: To characterize changes in emotion-processing neural networks associated with ketamine and rapid antidepressant response.

* Experiment 2.1: Neural changes in response to emotional faces associated with ketamine and rapid antidepressant response.

  o Hypothesis 2.1a: Ketamine, compared to midazolam, will be associated with reduced activation in the amygdala to sad compared to neutral faces. 2.1b: Antidepressant response, compared to non-response, will be specifically associated with changes in PFC/ACC function.
* Experiment 2.2: Neural changes during negative emotion regulation (cognitive reappraisal) associated with ketamine and rapid antidepressant response.

  * Hypothesis 2.2a: Ketamine, compared to midazolam, will be associated with reduced activation in the amygdala during negative emotion generation and enhanced PFC/ACC function during down-regulation of negative affect. 2.2b: Antidepressant response, compared to non-response, will be specifically associated with enhancement of PFC/ACC function.

Specific Aim 3 (Exploratory): To investigate functional and effective connectivity between emotion perception/generation neural systems and cognitive emotional regulation systems. Hypothesis 3: TRD compared to HC will be characterized by abnormal connectivity between PFC/ACC and amygdala, which will normalize with rapid antidepressant response.

The setting of research will be MSSM. All research participants will be recruited and screened through the Mood and Anxiety Disorders Program (MAP) (Director: Dan V. Iosifescu, M.D.) at MSSM. MAP is one of the major clinical research programs of the Department of Psychiatry, with research funding from NIH, the Department of Defense, NARSAD, and industry.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, 18-70 years of age;
* Participants must be free of any psychiatric condition (for the healthy volunteer group) or meet DSM-IV criteria for major depressive disorder, without psychotic features, based on the Structured Clinical Interview for DSM-IV TR Axis I Disorders (SCID);
* Participants have demonstrated inadequate response to a minimum of 1 adequate antidepressant treatment trial in current episode (e.g. TRD);
* Participants must be willing to undergo washout of psychotropic medications that he or she is taking;
* Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process.

Exclusion Criteria:

* Lifetime diagnosis of schizophrenia or any psychotic disorder, bipolar disorder, pervasive developmental disorders or mental retardation;
* Current diagnosis of obsessive-compulsive disorder (OCD), but not other anxiety disorders;
* Diagnosis of a substance use disorder within the past six months; all participants must have a negative urine toxicology test on the day of the fMRI, prior to the scan;
* Female participants who are pregnant, nursing, for may become pregnant;
* Any unstable medical illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease); endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease;
* Clinically significant abnormalities of laboratories, physical examination, or ECG;
* Participants judged to be at serious suicidal risk by the PI or another study-affiliated psychiatrist;
* Any contraindications to MRI, including pacemakers or metallic objects in the body.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research plan calls for the recruitment of adult human subjects with major depressive disorder (MDD) or healthy control (HC) volunteers over the 5-year grant period. All participants are required to be medically healthy as determined by medical history, physical examination, ECG, screening blood laboratory tests, urine analysis, and urine toxicology drug screen. Participants with MDD must have demonstrated inadequate therapeutic response to a minimum of one adequate antidepressant trial (e.g. TRD). MDD participants who meet this minimum TRD threshold will be eligible for the experiments in Aim 1.
  We recruit participants from several Mount Sinai-affiliated community hospitals (North General Hospital, Elmhurst), mental health associations (National Alliance for the Mentally Ill, Mood Disorders Support Group of New York), the Mood and Anxiety Disorders Program (MAP) Outpatient Clinic, the Mount Sinai Hospital outpatient psychiatry clinic, and from media/internet advertising.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2011-07-15 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale | baseline and 24hrs post fMRI scan
  The Montgomery-Asberg Depression Rating Scale (74) is a well-validated 10-item instrument with good ecological validity. It is used extensively in clinical research for the evaluation of depressive symptoms in adults, and is particularly sensitive to detecting change in symptoms. This scale serves as the primary depression-related behavioral rating for correlation with our neuroimaging data.

SECONDARY OUTCOMES:
Change in Clinician-Rated Inventory of Depressive Symptomatology (IDS-C30) | baseline and 24hrs post fMRI scan
  The 30-item Clinician-Rated Inventory of Depressive Symptomatology (IDS-C30) (75) is a clinician-rated instrument which includes all DSM-IV diagnostic criterion items for MDD as well as commonly associated symptoms such as anxiety, irritability, and melancholic and atypical symptom features.
Change in Brief Psychiatric Rating Scale and the Clinician-Administered Dissociative States Scale (CADSS) | baseline and 24hrs post fMRI scan
  Potential dissociative or other acute behavioral changes during the KET/MID infusions will be assessed using the Brief Psychiatric Rating Scale and the Clinician-Administered Dissociative States Scale (CADSS)

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States